Neurosciences Building, Department of Psychiatry, Warneford Hospital, Warneford Lane, Oxford, OX3 7 JX



Professor Catherine Harmer Principal Investigator +44 (0)1865 618326 catherine.harmer@psych.ox.ac.uk

Miss Catherine Hobbs, PhD Student University of Bath, c.hobbs@bath.ac.uk



The effect of acute citalopram on self-referential emotional processing and social cognition in healthy volunteers

NCT Number: Not yet available

Date: 30/09/19

## PARTICIPANT CONSENT FORM

CUREC Approval Reference: R64589/RE003

The effect of acute citalopram on self-referential emotional processing and social cognition in healthy volunteers

Purpose of Study: To investigate whether an acute dose of citalopram changes how the brain deals with emotional and social information about the self and others, in healthy participants.

| | | Please initial<br>each box |
|---|---|---|
| 1 | I confirm that I have read and understand the information sheet version 4.0 dated 10 <sup>th</sup> October 2019 for the above study. I have had the opportunity to consider the information carefully, ask questions and have had these questions answered satisfactorily. | |
| 2 | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, and without any adverse consequences or academic penalty. | |
| 3 | I have been advised about the potential risks associated with taking part in this research and have taken these into consideration before consenting to participate. | |
| 4 | I have been advised as to what I need to do for this research (especially with regard to drug intake) and I agree to follow the instructions given to me. | |
| 5 | To the best of my knowledge, I do not meet any of the exclusion criteria outlined in the information sheet for this research. If this changes at a later date during study participation, I agree to notify the researchers immediately. | |
| 6 | I understand that data collected during the study may be looked at by designated individuals from the University of Oxford and University of Bath. I give permission for these individuals to access my data. | |
| 7 | I understand that this study is a collaboration between the University of Oxford and University of Bath, and that data collected as part of this study may be used as part of a PhD thesis submitted to the University of Bath. | |
| 8 | I understand who will have access to personal data provided, how the data will be stored and what will happen to the data at the end of the project. | |
| 9 | I agree for data collected in this study to be shared with other researchers, including those working outside of the EU, to be used in other research studies. I understand that any data shared will be fully anonymised so that I cannot be identified. | |
| 10 | I understand that anonymised data will be made 'open data'. I understand that this means the anonymised data will be publicly available and may be used for purposes not related to this study, and it will not be possible to identify me from these data. | |
| 11 | I understand how this research will be written up and published. | |

| Name of | person taking consent | dd / mm / yyyy<br>Date | |
|---|---|---|---|
| Name of Participant | | dd / mm / yyyy<br>Date | Signature |
| 14 | I agree to take part in the | study | |
| 13 | I understand how to raise a concern or make a complaint. | | |
| 12 | I understand that this project has been reviewed by, and received ethics clearance through, the University of Oxford Central University Research Ethics Committee. | | |